CLINICAL TRIAL: NCT04640701
Title: Obesity in G60 Trauma Patients / Obesity in G60 Trauma Patients
Acronym: Obesity
Status: Completed | Type: Observational
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 046.TRA.2016.D
Record Dates: First submitted 2019-08-12; First posted 2020-11-23 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other:

SUMMARY:
Obesity is a national epidemic that affects all aspects of health care, including trauma care. According to the Centers for Disease Control and Prevention, 1% of US adults 20 years old and older are obese (body mass index [BMI], calculated as weight in kilograms divided by height in meters squared, > 30), and 69% are overweight (BMI > 25) (1, 2). Obesity is a major health concern because of its established relationship with serious medical diseases and increased likelihood of comorbid conditions (eg, diabetes mellitus, hyperlipidemia, heart disease, pulmonary disease) (3). As the number of obese adults continues to increase, the potential number of obese trauma patients with severe injury and complications will also increase (3). Management of prehospital and in-hospital trauma care, including complications associated with airway management, surgical procedures, and radiological imaging, of obese patients can be challenging. However, published reports on how obesity complicates hospital stays after trauma are conflicting (4, 5). Several studies have indicated that obese trauma patients are more likely than non-obese patients to have longer stays in the intensive care unit (ICU) and hospital, more days of mechanical ventilation, more complications, and comorbid conditions, and higher mortality (6,7,8). Other studies have indicated no differences between obese and nonobese patients in mortality, length of stay in the ICU and the hospital, duration of mechanical ventilation, complications, or comorbid conditions (9). Accordingly, the main aim of this study is to investigate and compare hospital course, clinical outcomes, disposition, and the cost of treatment between geriatric obese and non-obese patients hospitalized for treatment of traumatic injuries.

DETAILED DESCRIPTION:
This proposed research is a retrospective chart review to determine if trauma patients with different body mass indexes differed in hospital course, clinical outcomes, disposition, and the cost of treatment.

Records of trauma patients who were admitted to MHS between January1st 2006 and June 30th 2016 will be retrieved to review the clinical charts according to the investigator's inclusion and exclusion criteria.

Basic demographics and clinical outcomes parameters as noted above will be attained from the patient's medical records.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patient's ≥ 60 years of age.
2. Blunt and penetration injury.

Exclusion Criteria:

1. Pregnant and breastfeeding women.
2. Patients < 60 years of age

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Records of trauma patients who were admitted to MHS between January1st 2006 and June 30th 2016
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2016-07-12 (Actual); Primary Completion 2022-05-13 (Actual); Study Completion 2022-05-13 (Actual)

PRIMARY OUTCOMES:
Obesity's effect on the outcomes of geriatric trauma patients | January1st 2006 and June 30th 2016
  Type of Injury (length of stay)

SECONDARY OUTCOMES:
Body mass index | January1st 2006 and June 30th 2016
  Body mass index is calculated as weight in kilograms divided by height in meters squared, > 30). Weight (Kgs) & hight (cms) measured from subjects are combined to report BMI.
Length of stay | January1st 2006 and June 30th 2016
  measured in days
Injury severity score | January1st 2006 and June 30th 2016
  Injury severity score

CONTACTS AND LOCATIONS:
Overall Officials: Michael Truitt, M.D., Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- Methodist Dallas Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No